CLINICAL TRIAL: NCT03720366
Title: A Phase 1, 2-Part, Multicenter, Open-Label, 3-Arm Study to Determine the Effect of Enasidenib (CC-90007) on the Pharmacokinetics of Single Oral Doses of Caffeine, Dextromethorphan, Fexofenadine, Flurbiprofen, Midazolam, Omeprazole, Pioglitazone, and Rosuvastatin in Patients With Acute Myeloid Leukemia
Brief Title: A Study of Perpetrator Drug Interactions of Enasidenib in AML Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CC-90007-CP-004; U1111-1218-1974 (Registry Identifier: WHO)
Expanded Access: NCT03723057 (No longer available)
Record Dates: First submitted 2018-10-24; First posted 2018-10-25 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Enasidenib; CC-90007; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm 1: Administration of enasidenib and Arm 1 probes (Experimental): Part 1: Subjects will receive prescribed doses of Arm 1 probes on Day -1, followed by the first enasidenib dose on Day 1. Subjects will continue to take enasidenib once daily for 27 more days. On Day 28, subjects will receive the Arm 1 probes again together with the Day 28 dose of enasidenib. Part 2: the subjects continue to receive daily doses of enasidenib for the next 28 days (equivalent to a cycle). The subject will continue in subsequent cycles until the end of the study (28 months) or termination
  Interventions: Drug: enasidenib; Drug: Arm 1 probes
- Arm 2: Administration of enasidenib and Arm 2 probes (Experimental): Part 1: Subjects will receive prescribed doses of Arm 2 probes on Day -1, followed by the first enasidenib dose on Day 1. Subjects will continue to take enasidenib once daily for 27 more days. On Day 28, subjects will receive the Arm 2 probes again together with the Day 28 dose of enasidenib. Part 2: the subjects continue to receive daily doses of enasidenib for the next 28 days (equivalent to a cycle). The subject will continue in subsequent cycles until the end of the study (28 months) or termination
  Interventions: Drug: enasidenib; Drug: Arm 2 Probes
- Arm 3: Administration of Enasidenib and Arm 3 probes (Experimental): Part 1: Subjects will receive prescribed doses of Arm 3 probes on Day -1, followed by the first enasidenib dose on Day 1. Subjects will continue to take enasidenib once daily for 27 more days. On Day 28, subjects will receive the Arm 3 probes again together with the Day 28 dose of enasidenib. Part 2: the subjects continue to receive daily doses of enasidenib for the next 28 days (equivalent to a cycle). The subject will continue in subsequent cycles until the end of the study (28 months) or termination.
  Interventions: Drug: enasidenib; Drug: Arm 3 probes

INTERVENTIONS:
Drug: enasidenib — enasidenib
  Other Names: CC-90007, AG-221
Drug: Arm 1 probes — caffeine, dextromethorphan, flurbiprofen, midazolam, and omeprazole
  Arms: Arm 1: Administration of enasidenib and Arm 1 probes
Drug: Arm 2 Probes — digoxin and rosuvastatin
  Arms: Arm 2: Administration of enasidenib and Arm 2 probes
Drug: Arm 3 probes — pioglitazone
  Arms: Arm 3: Administration of Enasidenib and Arm 3 probes

SUMMARY:
This is a 2-part, open-label, interventional study conducted in approximately 42 subjects with AML harboring an IDH2 mutation.

The overall study is a 3-arm investigation of the PK effects of enasidenib at steady state on the probe compounds. (Part 1), followed by treatment continuation up to 28 months (Part 2).

Each arm utilizes different probe compounds; enrolls a separate cohort of approximately 14 subjects; and consists of 2 parts - investigation of the PK effects of enasidenib on the respective probe compound(s) (Part 1), followed by an enasidenib treatment extension (Part 2).

DETAILED DESCRIPTION:
Subjects can only be enrolled in one treatment arm. The probes (which are given twice) used in the study are approved for use in the countries where the study will be conducted. The probes in Arm 1 consist of single doses of caffeine (100mg), dextromethorphan (30 mg), flurbiprofen (50 mg), midazolam (0.03 mg/kg), and omeprazole (40 mg). Arm 2 probes consist of digoxin (0.25 mg), and rosuvastatin (10 mg). Arm 3 probe is pioglitazone (15 mg). Enasidenib is administered orally. All probes, except for midazolam, are administered orally. Midazolam will be administered intravenously.

In Part 1 (equivalent to Cycle 1), eligible subjects will receive the probes on Day -1, followed by the first dose of enasidenib on Day 1. Enasidenib will continue to be taken once daily for 28 days. Blood samples for pharmacokinetic analysis will be collected according to a set schedule. Subjects will receive the probes a second time on Day 28. Part 2 of the study begins the next day when the subject begins a second round of daily enasidenib doses (equivalent to Cycle 2). Safety assessment s and procedures consistent with AML standard of care will continue.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
2. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
3. Subject is ≥ 18 years of age at the time of signing the ICF.
4. Subject has either primary (ie, de novo) or secondary (associated with myelodysplastic syndrome [MDS], myeloproliferative neoplasms [MPN], or prior therapy with hematotoxins and/or radiation {ie, therapy-related disease}) AML according to the WHO classification.
5. Subject either:

   a. has received at least first line of AML therapy and any number of subsequent lines/regimens Note: For subjects having AML secondary to prior higher risk [Intermediate-2 or High risk according to the International Prognostic Scoring System] MDS treated with a hypomethylating agent [eg, azacitidine or decitabine], the hypomethylating therapy can be counted as a line/regimen if there is disease progression to AML during or shortly [eg, within 60 days] after the hypomethylating therapy.); or b. has never been treated for AML, but has declined standard of care chemotherapy.
6. Subject has the following disease status:

   1. Refractory to, or relapsed after first, second, or third line regimen of intensive therapy for AML (eg, the "7 + 3" protocol) with at least 5% leukemic blasts in bone marrow (the minimum number of treatment cycles of the intensive therapy is per the investigator's discretion); or
   2. Refractory to, or relapsed after first, second or third line low-intensity AML therapy (eg, low dose cytarabine (LDAC), azacitidine or decitabine) with at least 5% leukemic blasts in bone marrow after at least 2 treatment cycles; or
7. Subject has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
8. Subject has IDH2 gene mutations revealed by local testing in samples of bone marrow aspirate and/or peripheral blood, and confirmed positive in bone marrow aspirate and/or peripheral blood. Local testing may be performed during screening or within two months prior to screening with appropriate documentation and concurrence of Sponsor's Medical Monitor.
9. Subject has adequate organ function defined as:

   * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 3 x upper limit of normal (ULN), unless considered to be due to leukemic organ involvement, following review by the Sponsor's Medical monitor; and
   * Serum total bilirubin ≤ 1.5 x ULN, unless considered due to Gilbert's syndrome (eg, a gene mutation in UGT1A1) or leukemic organ involvement, following review by the Investigator and the Sponsor's Medical Monitor; and
   * Estimated glomerular filtration rate (GFR) > 30 mL/min based on the Modification of Diet in Renal Disease (MDRD) formula: GFR (mL/min/1.73 m2) = 175 × (serum creatinine)-1.154 × (Age)-0.203 × (0.742 if female) × (1.212 if African American)
10. Females of childbearing potential (FCBP)2 may participate, providing they meet the following conditions:

    * Agree to practice true abstinence from sexual intercourse or to use highly effective contraceptive methods (eg, combined [containing estrogen and progestogen] or progestogen-only associated with inhibition of ovulation, oral, injectable, intravaginal, patch, or implantable hormonal contraceptive; bilateral tubal occlusion; intra-uterine device; intrauterine hormone-releasing system; or male partner sterilization [note that vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success]) at screening and throughout the study, and for 4 months following the last study treatment; and
    * Have a negative serum β-subunit of human chorionic gonadotropin (β-hCG) pregnancy test (sensitivity of at least 25 mIU/mL) at screening; and
    * Have a negative serum β-hCG pregnancy test (sensitivity of at least 25 mIU/mL) within 72 hours prior to the start of study treatment in the Treatment Phase (note that the screening serum pregnancy test can be used as the test prior to the start of study treatment in the Treatment Phase if it is performed within the 72-hour timeframe).
11. Male subjects must agree to practice true abstinence from sexual intercourse or to the use of highly effective contraceptive methods with non-pregnant female partners of childbearing potential at screening and throughout the course of the study, and should avoid conception with their partners during the course of the study and for 4 months following the last study treatment.

Exclusion Criteria:

Presence of any of the following will exclude a subject from enrollment:

1. Subject is suspected or proven to have acute promyelocytic leukemia based on morphology, immunophenotype, molecular assay, or karyotype.
2. Subject has AML secondary to chronic myeloid leukemia (CML).
3. Subject has received a targeted agent against an IDH2 mutation.

   a. Prior treatment with an IDH2-targeted agent is acceptable if such treatment was interrupted for bone marrow or stem cell transplantation AND the patient was responsive to IDH2 treatment without progressive disease prior to transplantation.
4. Subject has received systemic anticancer therapy or radiotherapy < 14 days prior to the start of study treatment. Note that hydroxyurea is allowed prior to the start of study treatment for the control of leukocytosis (however, hydroxyurea should not be given within 72 hours prior to and after administration of azacitidine).
5. Subject has received non-cytotoxic or investigational agents < 14 days or 5 half-lives, whichever is longer, prior to the start of study treatment.
6. Subject has undergone hematopoietic stem cell transplantation (HSCT) within 60 days prior to the start of study treatment, or on immunosuppressive therapy post HSCT at the time of screening, or with clinically significant graft-versus-host disease (GVHD).

   a. The use of a stable dose of oral steroid post-HSCT and/or topical steroids for ongoing skin GVHD is permitted.
7. Subject has persistent, clinically significant non-hematologic toxicities from prior therapies.
8. Subject has or is suspected of having central nervous system (CNS) leukemia.

   a. Evaluation of cerebrospinal fluid is only required if CNS involvement by leukemia is suspected during screening.
9. Subject has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment).
10. Subject has immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation.
11. Subject has significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke; or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 6 months starting study treatment.

    1. The LVEF should be representative of the subject's daily status (ie, not collected during temporary disturbances such as sepsis, acute cardiac drug toxicity, acute pulmonary embolism, etc).
    2. An imaging-based assessment of left ventricular function may be collected at Investigator's discretion as part of screening if needed to resolve uncertainty regarding prior tests or current clinical status.
12. Subject is known seropositive or is infected with human immunodeficiency virus (HIV) or has active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV).
13. Subject is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally.
14. Subject has uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 100 mmHg).
15. Subject is a pregnant or lactating female.
16. Subject is known or suspected to have hypersensitivity to any of the components of PK probe compounds or study treatment.

    Note: A subject may be enrolled into an alternate arm of the study to which the subject does not have hypersensitivity if that alternate arm has not been filled, and if the alternate arm is available in the respective country. Subject is planning, or has reasonable probability, to violate the restrictions. Note in particular the medication restrictions.
17. Subject has QTc interval (ie, Fridericia's correction [QTcF]) ≥ 480 ms or other factors that increase the risk of QT prolongation or arrhythmic events (eg, heart failure, hypokalemia, family history of long QT interval syndrome) at screening. Reversible factors such as hypokalemia or hypomagnesemia may be corrected prior to dosing if the Investigator and Sponsor's Medical Monitor concur.
18. In conjunction with the restrictions, subject is taking the following CYP-sensitive substrate medications that have a narrow therapeutic range are excluded from the study unless the subject can be transferred to other medications at least 5 halflives prior to the start of study treatment: paclitaxel and docetaxel (CYP2C8), phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline, and tizanidine (CYP1A2).
19. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that places the subject at unacceptable risk or would prevent the subject from participating in the study.
20. Subject has any condition that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - AUC0-30 | Up to approximately 29 days
  Area under the probe plasma concentration-time curve calculated from time zero to 30 hours
Pharmacokinetics - Cmax | Up to approximately 29 days
  Observed maximum probe plasma concentration

SECONDARY OUTCOMES:
Pharmacokinetics - AUC0-∞ | Up to approximately 29 days
  Area under the probe plasma concentration time curve from time zero to infinity
Pharmacokinetics -t1/2,z | Up to approximately 29 days
  Terminal elimination half life for the probes
Pharmacokinetics - CL/F | Up to approximately 29 days
  Apparent clearance of probes from plasma
Pharmacokinetics - Vz/F | Up to approximately 29 days
  Apparent total volume of distribution of the probes, based on the terminal phase
Complete Response Rate | Up to approximately 28 months
  Measurement of tumor size reduction by a predefined amount over the defined time period
Adverse Events (AEs) | Up to approximately 28 months
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- Australia (7):
  - Local Institution - 103, Concord, New South Wales
  - Local Institution - 107, Adelaide, South Australia
  - Local Institution - 106, Clayton, Victoria
  - Local Institution - 102, Heidelberg, Victoria
  - Local Institution - 105, Nedlands, Western Australia
  - Local Institution - 101, Melbourne
  - Local Institution - 104, Waratah
- South Korea (3):
  - Local Institution - 203, Seoul
  - Local Institution - 202, Seoul
  - Local Institution - 201, Seoul

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/content/studyconnect/us/en/clinical-trials/NCT03720366.html